CLINICAL TRIAL: NCT02015442
Title: Effect of Eucaloric High and Low Sucrose Diets on Liver Fat in Healthy Adult Men With Liver Fat Levels Below 5%
Brief Title: Effect of Sucrose on Liver Fat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: SucroseLiver
Record Dates: First submitted 2013-12-13; First posted 2013-12-19 (Estimated); Results first posted 2019-11-14 (Actual); Last update posted 2019-11-14 (Actual); Status verified 2019-11

CONDITIONS: Healthy Volunteers
Keywords: Sucrose in diet
MeSH Terms: interventions — Sucrose

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High sucrose diet (Experimental): High sucrose diet for 7 days
  Interventions: Dietary Supplement: Sucrose
- Low sucrose diet (Experimental): Low sucrose diet for 7 days
  Interventions: Dietary Supplement: Sucrose

INTERVENTIONS:
Dietary Supplement: Sucrose

SUMMARY:
AIMS To determine the effect of high and low sucrose diets on liver fat in healthy adult men with liver fat levels below 5%

DETAILED DESCRIPTION:
DESIGN Randomized, cross-over design with two 7-day dietary interventions separated by a 4 week wash-out period. Dietary intervention will be based on iso-energetic substitution of sucrose for starch in a weight-maintaining diet. The two experimental conditions are: high sucrose diet at 25% of total energy intake (this is approximately the 95th percentile for UK intake of non-milk extrinsic sugars (NMES)); and low sucrose diet at 10% of total energy intake. Otherwise the macronutrient balance in both conditions will be based on UK average habitual intake.

POPULATION 10 healthy males aged between 20 and 40 years, with a BMI between 20-25kg/m2, with normal liver fat levels (<5%) and fasting plasma glucose and no evidence of insulin resistance will be recruited. No pre-existing morbidity including cardiac, hepatic or renal disease, history of diabetes, hypertension or hyperlipidemia. Usual physical activity of subjects to range from sedentary to a maximum of meeting the UK minimum activity recommendations (30 min moderate exercise 5 d/week). Habitual alcohol intake of less than 2 units per day.

TREATMENT Pre-intervention: Participants will be asked to record habitual dietary intake by completion of a 7-day food diary and be asked to wear an accelerometer armband to assess physical activity before each intervention week. Resting energy expenditure will also be assessed by indirect calorimetry.

7 day dietary interventions: Participants will be resident at the clinical research facility at Hammersmith Hospital during each intervention week for 5 out of the 7 days and all food will be provided at the facility. At the weekends, participants will have to leave the unit but food will be provided for those two days so that the diet can be continued at home.

At the start and end of each 7 day intervention: Weight, height and waist circumference will be taken; percentage liver fat and total and regional body composition will be measured by MRI. Fasting and post prandial plasma glucose, insulin and lipids will be measured and blood pressure.

ELIGIBILITY:
Inclusion Criteria:

Healthy men aged between 20 and 40 years with BMI between 20-25 kg/m2 and with normal liver fat levels (<5%), normal fasting glucose (less than 5.5mmol/l) and HbA1C less than 5.7% will be eligible to volunteer.

Exclusion Criteria:

* Type 1 diabetes, Type 2 diabetes, hypertension or hyperlipidaemia
* Gained or lost ≥ 3kg weight in the past three months
* Use of medication likely to interfere with metabolism, appetite regulation, glucose homeostasis and hormonal balance
* Regular consumer of sugar sweetened beverages
* Any chronic illness
* Cardiovascular, hepatic or renal disease
* Excess alcohol intake (>2 units per day)
* Exceeding UK minimum activity recommendation (30min moderate exercise 5d/wk)
* Current smokers (smoked within last 6 months)
* Any gastrointestinal disorder e.g. Crohn's disease, coeliac disease or irritable bowel syndrome
* A history of drug or alcohol abuse in the last 2 years
* Pancreatitis
* Unable to have MRI (eg. metallic or magnetic implants, claustrophobia)

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Frost, Principal Investigator — Imperial College London
Locations (1):
- NIHR/Wellcome Trust Imperial Clinical Research Facility, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- High Sucrose Diet Then Low Sucrose: High sucrose diet for 7 days, then low sucrose diet
- Low Sucrose Diet Then High Sucrose: Low sucrose diet for 7 days for first intervention, then high sucrose
Period: First Intervention (7 Days)
Arm/Group | High Sucrose Diet Then Low Sucrose | Low Sucrose Diet Then High Sucrose
Started | 5 | 4
Completed | 5 | 4
Not Completed | 0 | 0
Period: Wash-out (4 Weeks)
Arm/Group | High Sucrose Diet Then Low Sucrose | Low Sucrose Diet Then High Sucrose
Started | 5 | 4
Completed | 5 | 4
Not Completed | 0 | 0
Period: Second Intervention (7 Days)
Arm/Group | High Sucrose Diet Then Low Sucrose | Low Sucrose Diet Then High Sucrose
Started | 5 | 4
Completed | 5 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All participants, cross-over study
Arm/Group | All Participants
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 24 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 9

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in Liver Fat
Description: Liver fat was assessed by magnetic resonance spectrometry (MRS)
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | High Sucrose Diet | Low Sucrose Diet
Number analyzed (Participants) | 9 | 9
percentage of change | 1.9 (1.7) | 1.9 (1.9)
Statistical Analysis 1: Comparison: High Sucrose Diet; Baseline vs. treatment period; Test type: Superiority; p = 0.390, t-test, 2 sided
Statistical Analysis 2: Comparison: Low Sucrose Diet; Baseline vs treatment; Test type: Superiority; p = 0.204, t-test, 2 sided

2. Secondary Outcome: Changes in Fasting Triglyceride Levels
Description: Triglyceride levels assessed from plasma in fasting state
Time Frame: Baseline and 7 days
Measure: Mean (Standard Deviation); unit: mmol/l
Arm/Group | High Sucrose Diet | Low Sucrose Diet
Number analyzed (Participants) | 9 | 9
mmol/l
  Baseline | 0.9 (0.1) | 0.9 (0.4)
  7 days | 0.8 (0.3) | 0.7 (0.3)
Statistical Analysis 1: Comparison: Low Sucrose Diet; Baseline vs treatment; Test type: Superiority; p = 0.001, t-test, 2 sided — calculated
Statistical Analysis 2: Comparison: High Sucrose Diet; Baseline vs treatment; Test type: Superiority; p = 0.244, t-test, 2 sided
Statistical Analysis 3: Comparison: High Sucrose Diet vs Low Sucrose Diet; Test type: Superiority; p = 0.244, ANOVA

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | High Sucrose Diet | Low Sucrose Diet
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 0/9 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes